CLINICAL TRIAL: NCT04047641
Title: A Combination of Cladribine, Idarubicin, Cytarabine (CLIA) and Quizartinib for the Treatment of Patients With Newly Diagnosed or Relapsed/Refractory Acute Myeloid Leukemia (AML) and High-Risk Myelodysplastic Syndrome (MDS))
Brief Title: Cladribine, Idarubicin, Cytarabine, and Quizartinib in Treating Patients With Newly Diagnosed, Relapsed, or Refractory Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0153; NCI-2019-04730 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0153 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Blasts 20 Percent or More of Bone Marrow Nucleated Cells; High Risk Myelodysplastic Syndrome; Recurrent Acute Biphenotypic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent High Risk Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory High Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute | interventions — Cladribine; Cytarabine; Idarubicin; quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (idarubicin, cladribine, cytarabine, quizartinib) (Experimental): INDUCTION: Patients receive idarubicin Intravenous over 1 hours on days 1-3, cladribine intravenous over 1-2 hours on days 1-5, cytarabine Intravenous over 3 hours on days 1-5 (or days 1-3 for patients over age 60), and quizartinib by mouth daily on days 6-19. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR or CRp after Induction receive idarubicin Intravenous over 1 hours on days 1-2, cladribine Intravenous over 1-2 hours on days 1-3, cytarabine Intravenous over 3 hours on days 1-3, and quizartinib by mouth daily on days 4-28. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients who achieve CR or CRi/CRh after Consolidation receive quizartinib by mouth daily on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Idarubicin; Drug: Quizartinib

INTERVENTIONS:
Drug: Cladribine — Given Intravenous
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given Intravenous
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Idarubicin — Given Intravenous
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
Drug: Quizartinib — Given by mouth
  Other Names: AC-220; AC010220; AC220

SUMMARY:
This phase I/II trial studies the side effects and how well cladribine, idarubicin, cytarabine, and quizartinib work in treating patients with acute myeloid leukemia or high-risk myelodysplastic syndrome that is newly diagnosed, has come back (relapsed), or does not respond to treatment (refractory). Drugs used in chemotherapy, such as cladribine, idarubicin, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Quizartinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving quizartinib with cladribine, idarubicin, and cytarabine may help to control acute myeloid leukemia or high-risk myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of quizartinib (AC220) in combination with cladribine, idarubicin and cytarabine (ara-C) induction chemotherapy in newly diagnosed or relapsed/refractory patients with high-risk myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML).

II. To determine the safety of the combination.

SECONDARY OBJECTIVES:

I. To determine the overall survival and disease-free survival of patients treated with this combination.

II. To investigate correlations of response to this combination with a 81-gene panel of gene mutations both in patients with and without FLT3 mutations.

III. To identify individual treatment-resistant cell populations and their signaling state that may relate to clinical outcomes using CyTOF (cytometry by time of flight) and single cell sequencing.

OUTLINE:

INDUCTION: Patients receive idarubicin intravenously (IV) over 1 hour on days 1-3, cladribine IV over 1-2 hours on days 1-5, cytarabine IV over 2 hours on days 1-5 (or days 1-3 for patients over age 60), and quizartinib orally (PO) once daily (QD) on days 6-19. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients who achieve complete response (CR) or CR with incomplete platelet recovery (CRp) after Induction receive idarubicin IV over 1 hour on days 1-2, cladribine IV over 1-2 hours on days 1-3, cytarabine IV over 2 hours on days 1-3, and quizartinib PO QD on days 4-28. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients who achieve CR or CR with incomplete bone marrow recovery (CRi)/CR with partial hematologic recovery (CRh) after Consolidation receive quizartinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of

  * AML (World Health Organization [WHO] classification definition of >= 20% blasts, excluding Acute promyelocytic leukemia),
  * Acute biphenotypic leukemia or
  * High-risk MDS (> 10% bone marrow blasts)
* Frontline cohort: Patients aged 18 to 65 years
* Relapse cohort: Patients aged >=18 years old
* Patients may be newly diagnosed (Frontline cohort) or with prior therapy (Relapsed cohort) as follows:

  * For frontline cohort: Patients must be chemonaive, i.e., not have received any chemotherapy (except hydroxyurea [Hydrea] [no dose limit], tretinoin [atra] [no dose limit] or ara-C [one or two doses (max 2 gr/m^2 per dose)] for transient control of hyperleukocytosis) for AML or MDS. They may have received hypomethylating agents for prior MDS and transfusions, hematopoietic growth factors or vitamins. Temporary prior measures such as apheresis or Hydrea are allowed
  * For relapsed cohort: Patients with previously treated, relapsed or refractory AML, acute biphenotypic leukemia or high-risk MDS (> 10% bone marrow blasts)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Creatinine < 1.5 mg/dl
* Total bilirubin < 1.5 mg/dL, unless increase is due to hemolysis or congenital disorder
* Transaminases (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x upper limit of normal (ULN)
* Potassium, magnesium, and calcium (normalized for albumin) levels should be at least within institutional normal limits
* Ability to take oral medication
* Ability to understand and provide signed informed consent
* Baseline test of left ventricular ejection fraction >= 50%
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days
* WOCBP must use appropriate method(s) of contraception such as oral contraceptive pills (OCP), birth control shots, intrauterine device (IUD) etc. WOCBP should use an adequate method to avoid pregnancy until 30 days after the last dose of investigational drug. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as men with known azoospermia do not require contraception
* Patients with isolated extramedullary myeloid neoplasm will be eligible

Exclusion Criteria:

* Any coexisting medical condition that in the judgment of the treating physician is likely to interfere with study procedures or results
* Breastfeeding women
* Patients with current active malignancies or any remission for < 6 months, except patients with carcinoma in situ or with non-melanoma skin cancer who may be in remission for less than 6 months or have active disease
* Active clinically serious and uncontrolled infection. Patients with recent infections must have no temperature of >= 101 degrees Fahrenheit (F) for at least 48 hours (hrs) (before first dose, day 1)
* Patients with known significant impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of quizartinib
* Documented active central nervous system leukemia (patients with history of central nervous system [CNS] leukemia without active disease are allowed)
* Patients with a known confirmed diagnosis of human immunodeficiency virus (HIV) infection or active viral hepatitis
* Patients who have had any major surgical procedure within 14 days of day 1
* Impaired cardiac function including any of the following:

  * Screening electrocardiography (ECG) with a corrected QT (QTc) > 450 msec. The QTc interval will be calculated by Fridericia's correction factor (QTcF). The QTcF will be derived from the average QTcF in triplicate. Patients are excluded if they have QTcF >= 450. Subjects with prolonged QTcF interval in the setting of RBBB (right bundle branch block) may participate upon review and approval by the medical monitor. RBBB for patients' triplicate electrocardiograms (EKGs) can show false QTc prolongation; therefore, the cardiology collaborator for this study will manually review to provide an accurate reading of the QTc
  * Patients with congenital long QT syndrome
  * Sustained ventricular tachycardia requiring medical intervention
  * Any history of clinically significant ventricular fibrillation or torsades de pointes
  * Known history of second or third degree heart block (may be eligible if the patient currently has a pacemaker)
  * Heart rate of < 50/minute on pre-entry ECG
  * Left bundle branch block
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Patients with myocardial infarction or unstable angina within 6 months prior to starting study drug
  * Congestive heart failure (CHF) New York (NY) Heart Association class III or IV
  * Atrial fibrillation documented within 2 weeks prior to first dose of study drug
  * Known family history of congenital long QT syndrome
  * Patients who are actively taking a strong CYP3A4 inducing medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | From the date of start of treatment until event (resistance or relapse) or death, whichever occurred first, assessed up to 12 months
  Will be estimate using the Kaplan-Meier method for each patient cohort. In addition, efficacy EFS will be analyzed in the intent to treat (ITT) population per cohort.
Incidence of adverse events | Up to 12 months
  Defined as any clinically significant treatment-related grade 3 or greater non-hematologic toxicity. Patient toxicity data will be summarized using frequency and percentages, by type, grade and relationship to the study drugs.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 12 months
  Will be estimate using the Kaplan-Meier method for each patient cohort. In addition, efficacy OS will be analyzed in the ITT population per cohort.
Disease free survival (DFS) | Up to 12 months
  Will be estimate using the Kaplan-Meier method for each patient cohort. In addition, efficacy DFS will be analyzed in the ITT population per cohort.
Rate of response | Up to 12 months
  The rate of response will be estimated for each 28-gene panel of gene mutations for each patient cohort.
Change of FLT3 ligand level | Baseline up to 12 months
  Will also explore the change of FLT3 ligand level before and after treatment using summary statistics, by patient cohort and by other subgroups (i.e. age).
Change in the presence of other gene mutations | Baseline up to 12 months
  Will also explore the change in the presence of other gene mutations before and after treatment using summary statistics, by patient cohort and by other subgroups (i.e. age).

CONTACTS AND LOCATIONS:
Overall Officials: Musa Yilmaz, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org